CLINICAL TRIAL: NCT05334433
Title: Assessment of Child Behavior and Soft Tissue Reaction After Local Anesthetic Injection Using Needle Versus Needless Systems
Brief Title: Child Behavior After Local Anesthetic Injection Using Needless Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ayatallah Elsayed Mohamed Aly Bassiouny, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 3399444
Record Dates: First submitted 2022-04-05; First posted 2022-04-19 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Child Behavior
MeSH Terms: conditions — Child Behavior | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local anesthesia injection with the comfort in jet (Needless system) (Experimental): A needle-less injection approach will be used to administer the local anesthetic solution
  Interventions: Procedure: Local anesthesia injection
- Local anesthesia injection with needle injection (conventional technique). (Active Comparator): A conventional aspirating syringe fitted with 27-gauge long needles will be used to administer the local anesthetic solution.
  Interventions: Procedure: Local anesthesia injection

INTERVENTIONS:
Procedure: Local anesthesia injection — Local anesthesia administration

SUMMARY:
The aim of this study is to evaluate the effect of needless injection (comfort in ject) on child behavior and its effect on adjacent oral mucosa and soft tissue in children during local anesthesia injection in comparison to the conventional injection technique

ELIGIBILITY:
Inclusion Criteria:

* According to Wright's classification of child behavior, children are classified as cooperative or possibly cooperative.
* Children who are medically fit.
* Children who are capable of interacting on a mental level.
* Children between the ages of 6 to 8.
* First dental visit.

Exclusion Criteria:

* Children who struggle with behavioral control (uncooperative).
* Children who have a history of allergic reaction to local anesthetic drugs.
* Parental rejection for participation.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Child behavior (Feeling pain during injection) (Binary Yes/No) | During injection (Immediate) (No follow up)
  Pain perception during LA injection

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt, Cairo, Egypt